CLINICAL TRIAL: NCT03061097
Title: Randomized Controlled Trial of Autologous Microbiome Reconstitution to Prevent Colonization by Antibiotic rEsistant Bacteria
Brief Title: Autologous Fecal Microbiota Transplantation to Prevent Antibiotic Resistant Bacteria Colonization
Acronym: RACE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Microbiome Health Research Institute (Other)
Collaborators: Boston Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 200201691946
Record Dates: First submitted 2017-02-17; First posted 2017-02-23 (Actual); Results first posted 2020-12-07 (Actual); Last update posted 2021-05-05 (Actual); Status verified 2021-04

CONDITIONS: Antibiotic Resistant Strain
Keywords: Autologous Fecal Microbiota Transplantation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment (autologous fecal microbiota preparation) (Experimental): Participants randomized into the treatment arm will receive a single dose of autologous fecal microbiota preparation (auto-FMP) via enema following an infectious episode requiring antibiotics, with follow-up at day 3, 7, 28, and 6 months.
  Route of Administration: Enema Dosing Regimen: 125mL x 1 dose
  Interventions: Biological: Autologous fecal microbiota transplant (Auto-FMP Enema)
- Placebo (Placebo Comparator): Participants randomized to the placebo arm will receive a single dose of placebo FMT via enema following an infectious episode requiring antibiotics, with follow-up at day 3, 7, 28, and 6 months. The placebo enema preparation will be identical in appearance but will not contain human feces to prevent unmasking of the trial arms.
  Interventions: Other: Placebo Enema Preparation

INTERVENTIONS:
Biological: Autologous fecal microbiota transplant (Auto-FMP Enema) — FMT is the process by which processed donor microbiota material is transplanted into recipients. The aim is to reconstitute the normal intestinal microbial flora in recipients. In this study, the fecal microbiota preparation will be made from the participant's own stool and processed into an auto-FMP enema formulation.
  Arms: Treatment (autologous fecal microbiota preparation)
Other: Placebo Enema Preparation — The placebo enema preparation will be identical in appearance but will not contain human feces to prevent unmasking of the trial arms.
  Arms: Placebo

SUMMARY:
This study, a Randomized controlled trial of Autologous microbiome reconstitution to prevent Colonization by antibiotic rEsistant bacteria (RACE), seeks to investigate the safety, feasibility and the role of autologous fecal microbiota transplantation (FMT) for the prevention of antibiotic resistant bacteria (ARB) through microbiome restoration.

DETAILED DESCRIPTION:
Note: The Protocol and Statistical Analysis Plan document contains modifications from what is on file at the FDA to reflect redactions and formatting requirements for public posting on ClinicalTrials.gov

ELIGIBILITY:
Inclusion criteria for study enrollment

1. Long-term care residents associated with Boston University-Boston Medical Center nursing home consortium
2. Adults (18 years or older)

Inclusion criteria for randomization

1) Infection requiring antimicrobial treatment at the discretion of the treating physician

Exclusion criteria for study enrollment

1. Pregnant. Participants of childbearing age will undergo urine pregnancy testing
2. Participant or substitute decision maker unable to provide informed consent
3. Allergies to following ingredients generally recognized as safe: glycerol and sodium chloride
4. Current enrollment in hospice
5. Colostomy
6. Unable to adhere to protocol requirements
7. Any condition that the physician investigators deems unsafe, including other conditions or medications that the investigator determines puts the participant at greater risk from FMT
8. Recent travel (last six months) to high risk regions based on the International SOS Medical Risk Rating system
9. Recent exposure (last six months) to unsafe drinking water

Exclusion criteria for stool collection

Enrollment stool sample will be tested for ARBs and processed into autologous FMT treatment (if of qualifying size). Sample will not be collected if any of the following are true:

1. Oral or intravenous antibiotic exposure within the previous 6 weeks of stool collection date (topical antibiotics will be permitted)
2. Active gastrointestinal infection at stool collection
3. Fever at the time of stool collection
4. Currently ill or complaining of any of the following signs or symptoms of illness: fever, diarrhea, blood stools and/or vomiting
5. Participants with a history of gastrointestinal (GI) illness within the past 30 days prior to enrollment stool collection, that at the discretion of the site investigator could reasonably be caused by one of the following pathogens: 1) Vibrio spp. 2) Norovirus 3) Rotovirus 4) Adenovirus 5) Shiga toxin

Exclusion criteria for randomization

* Colonized with CRE (assessed by PCR or culture assay during enrollment phase)
* Colonized with VRE (assessed by PCR or culture assay during enrollment phase)
* Colonized with ESBL (assessed by PCR or culture assay during enrollment phase)
* Colonized with CDI (assessed by EIA assay on stool collected at enrollment phase)
* Treatment with antibiotics which are active against MRSA (i.e. vancomycin or linezolid) prior to randomization to FMT intervention or placebo.
* Stool culture positive for common enteric pathogens (Salmonella spp., Shigella spp., Campylobacter spp.)
* Participants who develop a GI illness with symptoms such as (but not limited to) vomiting or diarrhea within 30 days after collection of enrollment stool will be evaluated by the site investigator. If the site investigator determines that the symptoms were most likely caused by 1) Vibrio spp., 2) Norovirus, 3) Rotavirus, 4) Adenovirus, or 5) Shiga toxin, the enrollment stool will be sent out to test for these organisms. If the culture is positive for any of these organisms, the participant will be excluded from randomization
* Any condition that the physician investigators deems unsafe, including other conditions or medications that the investigator determines puts the participant at greater risk from FMT
* Participants who become severely immunocompromised, as defined by the investigator or treating physician, will be excluded prior to receiving intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2017-07-10 (Actual); Primary Completion 2018-12-19 (Actual); Study Completion 2019-06-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Majdi Osman, MD, MPH, Principal Investigator — Microbiome Health Research Institute, (d/b/a OpenBiome)
Locations (1):
- Boston University - Boston Medical Center nursing home consortium, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liu CK, Seo J, Pravodelov V, Frazier S, Guy M, Concilio K, Lau-Ng R, Brandeis G, Watson J, van der Velde J, Olesen SW, Budree S, Njenga M, Kassam Z, Osman M. Pilot study of autologous fecal microbiota transplants in nursing home residents: Feasibility and safety. Contemp Clin Trials Commun. 2022 Mar 7;27:100906. doi: 10.1016/j.conctc.2022.100906. eCollection 2022 Jun. PMID 35299780

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We enrolled 78 patients across four nursing homes from July 10, 2017 to June 30, 2018. Of these 78, a total of 33 individuals were able to provide a stool sample of sufficient quantity to undergo procedures required for preparation of autologous FMT. As specified in the protocol, only participants that had stool processed into autologous FMT and subsequently received a course of antibiotics will undergo randomization. Out of the 33 eligible participants, a total of 7 were ultimately randomized
Pre-assignment Details: Of the 7 randomized participants, 3 participants withdrew prior to administration of FMT. A total of 26 enrolled participants were withdrawn or discontinued prior to randomization for reasons including: enrollment in hospice care, passing away from age-related comorbidities, withdrawal of consent, and non-compliance. The remaining 45 enrolled participants were removed at study closure since they did not meet criteria for randomization at the time of closure.
Groups:
- Treatment (Autologous Fecal Microbiota Preparation): Participants randomized into the treatment arm will receive a single dose of autologous fecal microbiota preparation (auto-FMP) via enema following an infectious episode requiring antibiotics, with follow-up at day 3, 7, 28, and 6 months.
  Route of Administration: Enema Dosing Regimen: 125mL x 1 dose
  Autologous fecal microbiota transplant (Auto-FMP Enema): FMT is the process by which processed donor microbiota material is transplanted into recipients. The aim is to reconstitute the normal intestinal microbial flora in recipients. In this study, the fecal microbiota preparation will be made from the participant's own stool and processed into an auto-FMP enema formulation.
Period: Overall Study
Arm/Group | Treatment (Autologous Fecal Microbiota Preparation) | Placebo
Started | 4 | 3
Completed | 4 | 0
Not Completed | 0 | 3
Not completed — Withdrawal by Subject | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment (Autologous Fecal Microbiota Preparation) | Placebo | Total
Number analyzed (Participants) | 4 | 3 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 4 | 3 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 3 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 2 | 1 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (NIH Grade ≥2) at Day 7 After Randomization
Description: Number of participants with NIH Grade ≥2 adverse events at Day 7 after randomization.
Time Frame: Day 7 after randomization
Population: All three (3) participants assigned to placebo arm withdrew post-randomization but pre-treatment administration. One (1) participant was outside of treatment window following antibiotic exposure and therefore no longer eligible to receive the treatment. Two (2) participants withdrew consent prior to administration of the intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Autologous Fecal Microbiota Preparation) | Placebo
Number analyzed (Participants) | 4 | 0
Participants | 4 | 0

2. Secondary Outcome: Number of Patients With Clearance of Antibiotic Resistant Bacteria (ARB)
Description: Number of patients with clearance of ARB among patients colonized at Day 28 by Polymerase Chain Reaction (PCR) assay or culture-based assay. ARBs are: Carbapenem-resistant Enterobacteriaceae (CRE) by PCR or culture assay, Extended spectrum beta-lactamase (ESBL)-producing organisms by PCR or culture assay, Vancomycin-resistant enterococci (VRE) by PCR or culture assay, or Clostridium difficile by PCR
Time Frame: Day 28 after randomization
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Autologous Fecal Microbiota Preparation) | Placebo
Number analyzed (Participants) | 4 | 0
Participants | 0 | 0

3. Secondary Outcome: Number of Participants Who Develop Any ARB-associated Infections
Description: Number of participants who develop any ARB-associated infections following autologous FMT at Day 3, Day 7, Day 28, and Month 6
Time Frame: Day 3, Day 7, Day 28, Month 6
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Autologous Fecal Microbiota Preparation) | Placebo
Number analyzed (Participants) | 4 | 0
Participants | 0 | 0

4. Secondary Outcome: Number of Participants With NIH Grade ≥2 AEs at Day 28 and Month 6
Description: Number of participants with NIH Grade ≥2 adverse events (intermediate at Day 28 and long-term at Month 6) following autologous FMT.
Time Frame: Day 28, Month 6
Population: All three (3) participants assigned to placebo arm withdrew post-randomization but pre-treatment administration. One (1) participant was outside of treatment window following antibiotic exposure and therefore no longer eligible to receive the treatment. Two (2) participants withdrew consent prior to administration of the intervention. Note: the 1 participant who experienced Grade ≥2 adverse events experienced a total of two (2) adverse events by Month 6.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Autologous Fecal Microbiota Preparation) | Placebo
Number analyzed (Participants) | 4 | 0
Participants | 1 | 0

5. Other Pre Specified Outcome: Microbiome Disruption Indices (MDI) (16S rRNA Sequencing)
Description: MDI-community and MDI-species at baseline (pre-infection on the date of stool collection), post-antibiotics on the intervention/placebo date (Day 0, Day 3, Day 7, and Day 28)
Time Frame: Day 0, Day 3, Day 7, Day 28
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were collected for 6 months after randomization.
Description: For the placebo arm: All three (3) participants assigned to placebo arm withdrew post-randomization but pre-treatment administration. One (1) participant was outside of treatment window following antibiotic exposure and therefore no longer eligible to receive the treatment. Two (2) participants withdrew consent prior to administration of the intervention.
Arm/Group | Treatment (Autologous Fecal Microbiota Preparation) | Placebo
All-Cause Mortality (participants affected / at risk) | 2/4 | 0/0
Serious Adverse Events (participants affected / at risk) | 4/4 | 0/0
Other Adverse Events (participants affected / at risk) | 2/4 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Autologous Fecal Microbiota Preparation) (N=4) | Placebo (N=0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Death (General disorders) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Urinary tract infection (Renal and urinary disorders) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Autologous Fecal Microbiota Preparation) (N=4) | Placebo (N=0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hemorrhoids (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-09-17): https://cdn.clinicaltrials.gov/large-docs/97/NCT03061097/Prot_SAP_ICF_000.pdf